CLINICAL TRIAL: NCT00636025
Title: Anatomy of Subcutaneous Structures in Areas With and Without Cellulite Depressions by Magnetic Resonance Imaging
Brief Title: Cellulite and Magnetic Resonance Imaging
Status: Completed | Type: Observational
Sponsor: Doris Hexsel (Other)
Responsible Party: Sponsor-Investigator, Doris Hexsel, Dr. Doris Hexsel and Brazilan Center for Studies in Dermatology, Hexsel Dermatology Clinic
Organization: Hexsel Dermatology Clinic (Other)
Other Study IDs: 02-CBED07-04
Record Dates: First submitted 2008-03-11; First posted 2008-03-14 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Cellulitis
MeSH Terms: conditions — Cellulitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — None retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational

SUMMARY:
The purpose of this study is to compare the anatomy of subcutaneous structures in areas with and without cellulite on the buttocks of same subjects with a non invasive technique, Magnetic Resonance Imaging.

DETAILED DESCRIPTION:
A cross-sectional study was performed at a single center, in accordance with good clinical practice. Thirty women aged 18 to 50 were included in this study. An experienced dermatologist evaluated all of the subjects in a standing position, with relaxed gluteus muscles, using the CSS classification. An area with cellulite and another without cellulite on the contralateral buttock were selected. The area with cellulite had an evident depressed lesion, whereas the area without cellulite had no depressed or raised lesions, The selected cellulite depression was marked with a positive symbol using a skin marking pen.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent;
* Subjects agreeing to take part of all procedures of the study, after being fully informed on the objectives and nature of the investigations;
* Healthy female subjects over 18 years;
* Subjects presenting cellulite on the buttocks;
* Medical history and physical examination which, based on the investigator's opinion, do not prevent the patient from taking part in the study and use the product under investigation;
* Female subjects of childbearing age should present a negative urine pregnancy test and should be using an effective contraceptive method (3 months before the enrollment until the end of the study);
* Availability of the subject throughout the duration of the study (180 days);
* Subjects with sufficient schooling and awareness to enable them to cooperate to the degree required by this protocol.

Exclusion Criteria:

* Pregnant women or women intending to become pregnant during the study (next 3 months);
* Subjects participating in other clinical trials;
* Any condition that, in the opinion of the investigator, can compromise the evaluation of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Females patients with cellulite on the buttocks.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The presence and characteristics of the fibrous septa in areas with and without cellulite. | at baseline
  image from MRI

SECONDARY OUTCOMES:
The characteristics of the subcutaneous tissue in areas with and without cellulite. | at baseline
  image from MRI